CLINICAL TRIAL: NCT06070753
Title: A Prospective, Trial About Safety and Efficacy of Combined Treatment With Cerebrolysin in Acute Ischemic Hemispheric Stroke Patients Undergoing EndoVascular Treatment (EVT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Eichel, Dr. Eichel- Head of the Neurology Department, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0347-21-SZMC
Record Dates: First submitted 2023-06-11; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Acute Ischemic Stroke
Keywords: STROKE; Endovascular Thrombectomy
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — cerebrolysin; abrineurin

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants undergo EVT plus Cerebrolysin (Experimental): one group of patients should receive intravenous treatment with Cerebrolysin (30 ml/day) starting post EVT CT-Perfusion that will be performed not later than 3 hours from completion of EVT. Treatment will be continued for 10 consecutive days as one single daily infusion.
  Interventions: Drug: Cerebrolysin

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin, 30 ml/day as intravenous infusion, first infusion after completion of EVT. Daily infusion for 10 consecutive days.
  Other Names: Abrineurin

SUMMARY:
The goal of this clinical trial is investigate the efficacy of a neuro/vascular-protective treatment with the drug Cerebrolysin in patients with acute ischemic stroke. starting immediately after completion of a EVT therapy.

The main question the study aims to answer is: If a 10 days treatment with the neuro/vascularprotective drug Cerebrolysin (30 ml/day as intravenous infusion) is able to increase the overall outcome of EVT therapy? Participants will receive intravenous treatment with Cerebrolysin (30 ml/day) starting immediately after thrombolytic therapy and being continued for 10 consecutive days as one single daily infusion. The modified Rankin Scale (mRS) 90 days after onset of symptoms will be investigated, but also the improvement in other ratings as well as the time course of the improvement.

In addition to the clinical outcome measures the study will assess neuroimaging perfusion CT-Perfusion parameters to evaluate possible direct improvement in microcirculation that might be an additional mechanism of action of cerebrolysin.

CT-Perfusion being done immediately after EVT will provide ability to stratify the data according to non-favorable CT-Perfusion parameters after EVT versus favoravle.

DETAILED DESCRIPTION:
9.1. Overall Study Design and Plan-Description

The study will be conducted as a single center, trial. In patients with AIS after EVT, according to the consensus guidelines, the study drug (Cerebrolysin) will be administered as IV-infusion over 30 minutes. First treatment will be administered up to 3 hours after completion of the EVT intervention.. First treatment will be given after a post EVT CT-Perfusion was performed. The treatment with Cerebrolysin will be repeated until day 10 as a single daily infusion. Patients may be inpatients as long as deemed necessary by the principal investigator. The observation period will last 9 (±14) month days after the administration of study medication. Patients recruited but not treated with the study drug due to various reasons or who do not receive the total dose of study medication will also be observed for 9 month if they survive.

The study is planned to be started in October 2023 (first patient in) and should be finished by June 2024.

The study will be conducted at the Shaare Zedek Medical Center. Treatments must be performed by a physician specialized in neurological care.

9.2. Discussion of Study Design, Including the Choice of Control Groups

9.2.1. Randomization No Randomization will be needed. 9.2.2. Treatment groups

Cerebrolysin has a neuro/vascularprotective mode of action. It is assumed, based on preclinical data and on first findings from clinical studies, that treatment with Cerebrolysin may be able to prevent neuronal death after brain ischemia. Therefore one group of patients should receive intravenous treatment with Cerebrolysin (30 ml/day) starting after post EVT CT-Perfusion that will be performed not later than 3 hours from completion of EVT. Treatment will be continued for 10 consecutive days as one single daily infusion.

9.2.3. Efficacy assessment tools The main goal of this study is to assess efficacy. Potential effects of EVT will be evaluated by using the mRS score at day 90 (primary endpoint). For the list of further endpoints see chapter 9.5.1.1.2. Secondary efficacy parameters.

Efficacy parameters: The NIH Stroke Scale will be performed at baseline, 1 hours (after Drug administration), 2 hours (after), 24 hours (after), Day 5, Day 10, on Day 7 and/or discharge, 30 days, 90 days and 9 month after the start of treatment. The Modified Rankin Scale on Day 7 and/or discharge, 30 days, 90 days and 9 month. All investigations should be done by an MRS and NIHSS certified investigator. Length of stay in hospital in both groups will be assessed as well. The patient termination record will be performed at 9 month or if a patient decides to withdraw the consent for further remaining in the study. Additional to clinical efficacy parameters the all outcomes measurements will be stratified by post-EVT CT-Perfusions measurements with a favourable and ubfavorable CT-Perfusion group.

9.2.4. Duration of the treatment

No later the 3 hours post EVT patient is brought to the MRI for ASLPV measurement the first infusion of the study medication (Cerebrolysin/Placebo) is administered as an IV-infusion over a time period of 30 min while patient is undergoing further MRI imaging with another ASLPV measurement at the end of the treatment . The treatment with Cerebrolysin will be repeated until day 10 as a single daily infusion every 24 +/- 2h. Patients may be inpatients as long as deemed necessary by the principal investigator. The observation period will last 9 month after the admission to the hospital with symptoms of acute ischemic stroke, qualifying for the study. Patients randomized, but not treated with Cerebrolysin because of any given reason or who do not receive the total dose of study medication, will also be observed for 9 month if they survive.

9.2.5. Choice of Cerebrolysin dosages

A dosage of 30 ml of Cerebrolysin per day over a period of 10 days has been chosen based on the results of previous preliminary trials in various indications, proofing to be the most efficacious dose. This finding is in compliance with data from preclinical studies, showing highest degree of neuroprotection in comparable dose ranges. An early start of treatment after EVT should ensure maximum rescue of neurons in the acute stage due to the neuro/vasculareprotective mode of action. The prolongation of the therapy over ten days should help to induce repair processes due to the neurotrophic properties of Cerebrolysin inducing neuronal sprouting reaction and maybe even proliferation and differentiation of neuronal progenitor cells.

Drug profile Cerebrolysin is a brain derived peptide preparation produced by a standardised enzymatic breakdown of lipid-free brain proteins. It consists of approximately 25% of low molecular weight peptides, based on the total nitrogen content, stabilised with amino acids. The drug is free from proteins, lipids and antigens and is administered by intravenous infusion (Summary, see also Investigator Brochure).

Qualitative and quantitative composition

1. ml contains 215.2 mg porcine brain derived peptide preparation (Cerebrolysin concentrate) in aqueous solution.

   Pharmaceutical form Cerebrolysin is a solution for injection/concentrate for solution for infusion. The vials ready for infusion have to be stored at room temperature (not over 25°C) in a dry place away from light.

   9.2.6. Treatment period

   The study drug will be administered first time as intravenous-infusion (30 ml of Cerebrolysin in a total volume of 100 ml, diluted with physiological saline) over 30 minutes not later the 3 hours after EVTand after psot EVT CT-Perfusion imaging..

   Treatment will be repeated on further 9 consecutive days (total of 10 administrations) if possible always as a morning dose. Patients may be inpatients as long as deemed necessary by the principal investigator. Patients are coming to hospital for all visits up to Day 10, if they can be discharged from hospital earlier.

   The observation period will last 9 month (±1week) after the first administration of study medication. Patients randomized but not treated with Cerebrolysin or who do not receive the total treatment course of study medication will also be observed for 9 month.

   9.3. SELECTION OF STUDY POPULATION Patients presenting with acute stroke ischemic stroke and being treated by successfully by EVT will be enrolled.

   9.3.1. Inclusion criteria

   To be eligible, the following inclusion conditions must be met:
   * Female or male inpatients.
   * Age: ≥18 years.
   * MRS ≤2
   * Clinical diagnosis of ischemic stroke eligible for EVT.
   * No Contraindication to perform CT-Perfusion.A) Patient is willing to participate voluntarily and to sign a written patient informed consent. Informed consent will be obtained from each patient or the legally authorised representative or two independent physicians, according to the regulatory and legal requirements of israel.
   * B) Patients who are unable to sign but who are able to understand the meaning of participation in the study may give an oral / physical witnessed informed consent. These patients have to make clear undoubtfully that they are willing to participate voluntarily and must be able to understand an explanation of the contents of the information sheet. The investigator and an independent witness have to sign the informed consent before any study specific procedures are performed. As soon as the medical condition of the patient is improving, obtaining of a written informed consent from the patient has to be achieved.

   C) Patients who are incapable of giving consent may be included as well. These patients have to sign a written consent as soon as they are able to understand the meaning of participating in the study and are able to sign. Two independent physicians not involved in the study have to sign the informed consent before any study specific procedures are performed. As soon as the patient is recovering, obtaining of oral, physical or written informed consent has to be achieved.

   If patients are not willing to stay in the study they have to be asked if data obtained so far can be used. This has to be documented on a separate form.

   • Willingness and ability to comply with the protocol after consenting.

   All inclusion criteria and none of the exclusion criteria listed below have to be achieved to include a patient.

   9.3.2. Exclusion criteria

   Brain Imaging • Evidence of intracranial haemorrhage (ICH) on the CT-scan

   General
   * Participation in another therapeutic clinical trial 3 months before baseline
   * Female patient of childbearing age must not be pregnant as proved by Beta-HGB negative testing.

   Medical • Platelet count of below 100x103/mm3
   * Blood glucose <50
   * Known haemorrhagic diathesis
   * Manifest or recent severe or dangerous bleeding
   * Known bacterial endocarditis, pericarditis
   * Acute pancreatitis
   * Documented ulcerative gastrointestinal disease during the last 3 months, oesophageal varices, arterial-aneurysm, arterial/venous malformation
   * Neoplasm with increased bleeding risk
   * Severe liver disease, including hepatic failure, cirrhosis, portal hypertension, oesaphageal varices) and active hepatitis
   * Major surgery or significant trauma in past 3 months
   * Multiple serious drug allergies
   * Hypersensitivity or allergy to one of the components of the drug
   * Severe renal impairment

   Psychiatric • Chronic intoxication or chronic substance use disorder with pharmaceuticals, drugs, alcohol or industrial poisons

   Neurological

   • Epilepsy

   • Symptoms suggestive of subarachnoid haemorrhage, even if the CT-scan is normal

   • Known history of or suspected intracranial haemorrhage

   • Suspected subarachnoid haemorrhage or condition after subarachnoid hemorrhage from aneurysm

   • Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)

   • Haemorrhagic retinopathy, e.g. in diabetes (vision disturbances may indicate haemorrhagic retinopathy)

   9.3.3. Removal of subjects from treatment or assessment

   Each patient may terminate the study prematurely without giving any reason. If possible, the patient should discuss her/his decision with the investigator. The investigator may terminate the administration of study drug prematurely for any medical reason. Reason as well as date and time of termination have to be documented. Each of these patients must be followed up for 9 month if possible. Drop-outs and withdrawals will not be replaced.

   Patients may be withdrawn from the study by the investigator at any time for any of the following reasons:

   • The patient does not follow the invitation to the scheduled clinical visits within 7 days from the scheduled visit.

   • When there are doubts that they comply with intake of study medication and use of allowed concomitant medication.
   * Whenever the patients are moving to a new location too far away from the hospital so that further participation in the study becomes questionable.

   Absolute withdrawal criteria for this study are:
   * Safety/efficacy reasons in the best interests of the patient.
   * Patient withdraws his/her consent.
   * Events that would obscure treatment effects, such as second stroke, epilepsy.
   * Malignancies developed/diagnosed during the trial
   * The randomisation code is broken.
   * The patient is lost to follow up.

   Conditions developing during the course of the study listed in the exclusion criteria as well as protocol deviations do not necessarily lead to the patient's withdrawal but should be properly documented.

   Patients who are withdrawn from the study due to AEs will be treated according to standard clinical strategies and will be followed up until they are resolved or stabilised or until a plausible explanation for the cause of the event has been found. All pertinent information concerning the outcome of the Adverse Event will be documented in the case report form.

   In accordance with the informed consent and the Declaration of Helsinki, the patient may discontinue the study at any time without any penalty or loss of benefits to which the patient is otherwise entitled. Reason(s) for a premature termination should be documented in the case report form. The final examination should be performed in such cases for safety reasons.

   Patients discontinuing the study must be fully documented up to the time of discontinuation. Both the discontinuation of the treatment and the reason why the treatment was prematurely terminated must be recorded in the case report form. In addition, time, date and circumstances should also be stated.

   9.3.4. Premature termination or suspension of the study The clinical study can be prematurely terminated or suspended by the PI after reassessing the risks of the study.

   A premature termination may be necessary for the following reasons:
   * The incidence of Adverse Events constitutes a potential health hazard.
   * New scientific data on the investigational product do not justify a continuation of the clinical study.
   * Serious and/or persistent non-adherence to the protocol, GCP and/or applicable regulatory requirements by an investigator/institution.

   Furthermore, the PI has the right to terminate the study for any reason at any time. If the study is prematurely terminated or suspended, the investigator has to inform the patients and to assure appropriate follow-up for the patients. The PI should promptly inform the investigators/institutions and the regulatory authority(ies) of the termination or suspension and the reason(s) for them. The IRB/IEC should also be informed promptly and provided the reason(s) for the termination or suspension by the sponsor or by the investigator/institution, as specified by the applicable regulatory requirement(s).

   9.4. TREATMENTS

   9.4.1. Treatments administered The study drug Cerebrolysin will be administered as a single daily dose of 30 ml diluted with physiological saline to a total volume of 100 ml as an intravenous infusion over a time period of 30 min..

   9.4.2. Identity of the investigational product Intravenous Study Medication (Cerebrolysin or Placebo) The IV study medication is packaged in amber glass vials containing 100 ml ready-to-use infusion solution. This infusion solution will either contain 30 ml Cerebrolysin + 70 ml physiological saline (0.9% NaCl) or 100 ml physiological saline (0.9% NaCl) only according to the randomisation plan. Batch number and expiry date are documented in the Trial Master File.

   Study medication will be infused daily for 10 consecutive days, giving a total of 10 infusions. The first infusion shall start not later than 3 hours after completion of EVT (Visit 1B). Infusions will take place only at the clinical facility.

   For each patient, 10 plus 2 replacement vials of study medication will be provided. The 10 vials will packaged in a carton; the two replacement vials per patient will be packaged in two separate carton boxes with the appropriate labeling.

   Preparation of study medication The study medication is supplied as a ready-to-use product for Israel. No special preparation of the study medication is required there.. Sterile NaCl (70 ml) will be available in amber 100 ml glass vials. 30 ml Cerebrolysin (3 x 10 ml) or 3 x 10 ml Placebo will be added under aseptic conditions up to a final volume of 100 ml. In addition, supplies for the administration of the infusions including IV lines, butterfly needles, adhesive tapes and alcohol swabs will be provided.

   THE STUDY MEDICATION WILL BE LABELLED AS FOLLOWS:

   Intravenous Study Medication (Cerebrolysin)

   VIALS:

   BOXES AND OUTER CARTON:

   Other information will be included as per specific country requirements.

   The final label of the study medication will be defined country specific according to ICH-GCP as well as local requirements and will be filed in the investigator and trial master file.

   BOXES: REPLACEMENT VIALS

   9.4.3. Method of assigning subjects to treatment groups

   Not needed everybody is receiving Cerebrolysin. 9.4.4. Selection of doses in the study The study will be conducted as a fixed-dose study in which one group of patients will receive 30 ml Cerebrolysin diluted with 70 ml physiological saline to a total volume of 100 ml. The other group will receive 100 ml of physiological saline as Placebo as a once daily infusion over a time period of 30 min. Start time and end of the infusion have to be recorded in the CRF.

   A dosage of 30 ml (OD) of Cerebrolysin is considered to be effective for the treatment of mild to moderately severe Alzheimer's Disease as shown in clinical studies and it has also shown efficacy in preliminary stroke trials. From previous experience it is suggested that this dosage should exert favourable clinical effects. This trial should also provide data on safety and tolerability of Cerebrolysin used immediately after thrombolytic therapy in patients suffering from acute ischemic stroke. Therefore the dosages should be maintained over the whole study period.

   All patients will receive a total of 10 infusions of study medication during the study on consecutive days.

   9.4.5. Selection and timing of dose for each subject The study will be conducted as a fixed-dose study in which Cerebrolysin-treated patients will receive a once daily dosage of 30 ml of the study medication, diluted with 70 ml of physiological saline to a total volume of 100 ml as intravenous infusion over a time period of

30 minutes. Dosage adjustments are not permitted. Patients experiencing dose limiting Adverse Events must be withdrawn from the study.

The first dosage will be applied immediately after the 1 hour rating which will be done after the end of the EVT therapy. Regardless the exact time of the first application, the next infusion of the study medication should be done on the next morning, between 07:00 and 10:00 a.m. All other treatments should be applied at approximately the same time of day within a time window of +/-2 hours.

9.4.6. Administration of study medication A butterfly needle will be inserted in a peripheral vein. Active treatment or Placebo will be infused intravenously over a period of approximately 30 minutes. The time of infusion will be recorded. The infusion will take place at approximately the same time every day within a time window of +/-2 hours.

The infusion will only be administered, if the patient does have vital sign values within the following ranges:

Supine BP systolic <200 mm Hg Diastolic <110 mm Hg Heart Rate 45-110/min. Body Temperature <38.0°C Respiratory Rate 10-30/min.

If one of the parameters is above the upper or below the lower limit, the nurse should wait for a few minutes and recheck the parameter. If the second measurement is within the limits, the infusion can be administered. Vital signs will be rechecked and recorded at the conclusion of the infusion. If a patient misses an infusion it may be added at the end of the treatment period to give a total of 10 infusions for that patient. A patient should not miss more than one consecutive infusion during the whole treatment period.

9.4.7. Blinding Not needed all patients are receiving Cerebrolysin. Blind will only exist in term of results of Post-EVT CTP results.

9.4.8. Prior and concomitant therapy

Additional thrombolytic medication (e.g. urokinase or streptokinase) is forbidden.

Brain protective drugs (e.g. brain specific calcium channel blockers or nootropics) are prohibited during the whole study period.

Other drug therapy may be given according to patient needs. Osmotic agents (mannitol, glycerol) may be given, if the intracranial pressure is increased.

Medication administered 48 hours prior to entry into the study must be recorded on the appropriate CRF page.

All concomitant medication must be recorded (date of onset, highest total daily dose, stop date and route of administration). If usage is prophylactic, this must be indicated on the respective CRF page.

9.4.9. Treatment compliance and drug accountability

The study medication (Cerebrolysin/Placebo) will be administered as single daily IV-infusion by the investigator or Coinvestigator for 10 consecutive days, starting not later than 3 hours after completion of EVT and after post EVT CT-Perfusion imaging. Compliance issues therefore do not play a role.

Drug supplies, which will be provided by the PI, must be kept in a secure, limited access storage area under the storage conditions defined by the sponsor. Where necessary, a temperature log must be maintained to ensure that the drug supplies are stored at the correct temperature.

The investigator and/or pharmacist must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each subject and the return to the sponsor or alternative disposition of unused products. These records will include dates, quantities, batch/serial numbers, expiry dates (if applicable) and the unique code numbers assigned to the investigational products and trial subjects. Investigators will maintain records that document adequately that the subjects were provided the doses specified by the protocol and reconcile all investigational products received from the sponsor.

A drug supply inspection for inventory purposes and to ensure proper storage will be conducted at regular intervals throughout the study.

9.5. EFFICACY AND SAFETY VARIABLES

9.5.1. Efficacy and safety measurements assessed and flow chart A patient may be enrolled into the study after giving his/her informed consent (or deferred in exceptional circumstances, according to national regulatory and legal requirements) when entering the clinic with acute stroke symptoms and after successful EVT treatment.

All inclusion and exclusion criteria have to be checked prior to administration of the test dose of study medication. The visit 1 is divided into three sub-visits. Five visits will be conducted during the study.

At visit 1A (baseline) the documentation of demographics, medical history, clinical lab, physical examination, vital signs, resting 12-lead ECG, concomitant therapy, NIH Stroke Scale at admission to hospital, modified Rankin Scale prior to ischemic stroke event, documentation of Adverse Events, pregnancy test (if appropriate).

The patient's informed consent is mandatory before these investigations are performed or can be deferred in exceptional circumstances, according to IRB of SZMC.

At visit 1B (not later than 3 hours after EVTand after post EVT CT-Perfusion), Infusion of the trial medication. At the end of the infusion Heart rate and blood pressure will be measured every 15 minutes until Hour 2.

At visit 1C (1 hour after the start of infusion of Cerebrolysin/Placebo), the NIH Stroke Scale will be performed, the documentation of Adverse Events and concomitant medication will be done. Heart rate and blood pressure will be measured every 30 minutes until Hour 6, then every hour until Hour 24.

At visit 2 (Day 5), heart rate and blood pressure will be measured. The documentation of Adverse Events and concomitant medication will be done. The NIH Stroke Scale and the modified Rankin Scale will be performed.

At visit 3 (Day 10), heart rate and blood pressure will be measured. The documentation of Adverse Events and concomitant medication will be done. The NIH Stroke Scale and the modified Rankin Scale will be performed.

At visit 4 (Day 7 and/or discharge), heart rate and blood pressure will be measured. The documentation of Adverse Events and concomitant medication will be done. The NIH Stroke Scale , GDS, MoCA, SF36 and the modified Rankin Scale will be performed.

At visit 5 (Day 30), heart rate and blood pressure will be measured. The documentation of Adverse Events and of concomitant medication will be done. The NIH Stroke Scale, GDS, MoCA, SF36 and the modified Rankin Scale will be performed.

At visit 6 (Day 90), the documentation of Adverse Events and concomitant medication will be done. Vital signs, the NIH Stroke Scale, GDS, MoCA, SF36 and the modified Rankin Scale will be performed.

At visit 7 (9 month +/- 7 days), heart rate and blood pressure will be measured. The documentation of Adverse Events, concomitant medication and a clinical lab will be done. The NIH Stroke Scale, GDS, MoCA, SF36 and the modified Rankin Scale will be performed. A physical examination takes place. The patient's termination record will be filled in. Length of stay in hospital in both groups will be assessed as well.

For visit 1A (D1) there is no time window (must take place within 30 after EVT) For visit 1B a window of ±10 minutes is acceptable. For visit 1C a window of ±15 minutes is acceptable. For visit 2 (D5) a window of ±1 hour is acceptable.

For visit 3 (D10) a window of ±1 hour is acceptable. For visit 4 (D7/discharge) a window of ±1 hour is acceptable. For visit 5 (D30), a window of ±1 day is acceptable For visit 6 (D90), a window of ±2 days is acceptable For visit 7 (9 month), a window of ±7 days is acceptable

In this study 5 visits are planned. The last examination takes place at 9 motnh ±7 days. BP/HR:

For assessing safety, blood pressure and heart rate are to be measured supine at baseline (prior to administration of trial medication). Further BP/HR monitoring will take place in the following order: every 15 minutes until Hour 2 (i.e. after 15, 30, 45, 60, 75, 90, 105, 120 minutes starting the infusion of Alteplase), every 30 minutes until Hour 6 (i.e. 150, 180, 210, 240, 270, 300, 330, 360 minutes) and every hour until Hour 24. Thereafter up to Day 10 BP and HR have to be recorded twice daily, before and after each Cerebrolysin-infusion (supine after 5 minutes rest).

ECG: Resting 12 lead-ECG readings are to be taken at baseline and on Day 10.

Adverse Events (AE):

AEs (free reporting by the patient after having been asked by the physician every day during the hospital stay) will be documented until hospital discharge (date and time of onset, date of last occurrence, intensity, etc.). From hospital discharge up to Day 90 only serious AEs will be reported.

Efficacy parameters:

The NIH Stroke Scale will be performed at baseline and 1 hour (after Drug administration), 2 hours (after), 24 hours (after), Day 5, Day 10 and Day 7/discharge, 30, 90 and 9 month. The Modified Rankin Scale will be performed on baseline, Day 7/discharge, 30, 90 and 9 month.

MoCA will be performed on Day 7/discharge, 30, 90 and 9 month. GDS will be performed on Day 7/discharge, 30, 90 and 9 month. The SF36 will be assessed on day 90 and after 9 month.

Length of stay in hospital in both groups will be assessed as well. The patient termination record will be filled in on 9 month.

9.5.1.1. Efficacy assessments

To ensure the sensitivity and reliability of efficacy assessment always the same rater for a given instrument should assess the status of a given patient at all visits.

9.5.1.1.1. Primary efficacy parameters

Modified Rankin Scale mRS score at Day 90 Rankin index: 7-point ordinal categorical scale: 0 - Full recovery to 6 - Death.

Possible to reduce to binary form (Success/Failure). χ2 analysis of difference in success rates between groups.

5 possible binary splits and 5 possible analyses. Parameter will be an overall measure of the advantage of the Treatment over Control accounting for each category.

Interpreted as a symptomatic improvement in the probabilities of desirable outcomes (MRS ≤2) at the expense of the undesirable outcomes(MRS ≥3).

9.5.1.1.2. Secondary efficacy parameters Modified Rankin Scale mRS score at Day7/discharge and day 30 Rankin index: 7-point ordinal categorical scale: 0 - Full recovery to 6 - Death.

Possible to reduce to binary form (Success/Failure). χ2 analysis of difference in success rates between groups.

5 possible binary splits and 5 possible analyses. Parameter will be an overall measure of the advantage of the Treatment over Control accounting for each category.

Interpreted as a symptomatic improvement in the probabilities of desirable outcomes (MRS ≤2) at the expense of the undesirable outcomes(MRS ≥3).

National Institute of Health Stroke Scale NIHSS 7/discharge 30,90 days and 9 month Difference between treatment groups regarding NIHSS <8, χ2 analysis of difference in success rates between groups.

MOCA 7/discharge,30,90 days and 9 month Difference between treatment groups regarding median MOCA, χ2 analysis of difference between groups.

Geriatric Depression Scale GDRS 7/discharge,30,90 days and 9 month Difference between treatment groups regarding median GDRS, χ2 analysis of difference between groups.

SF36 90 days and 9 month Difference between treatment groups regarding median SF36, χ2 analysis of difference in between groups.

mRS- Stratified by favorable versus unfavorable post ECT CT Perfusion measruements

9.5.1.1.3. Diagnostic variables NA

9.5.2. Appropriateness of measurements Cerebrolysin has already shown efficacy in smaller studies using the same or at least similar rating scales. The rating scales used in the study reflect state of the art as also applied in many other drug studies in stroke.

The scales are relevant to document the neurological status of the patient at any given time point of the trial.

The selection was also supported by the fact that these scales have been used for the thrombolytic studies as well, so a direct comparison to the results of these studies will be possible, to get additional information about a possible benefit of the adjuvant therapy with Cerebrolysin on outcome of patients suffering from acute ischemic stroke.

9.5.3. Efficacy variables 9.5.3.1. Primary efficacy variable(s)

Modified Rankin Scale: a complete description of the scale is given in Appendix 11.4.

9.5.3.2. Secondary efficacy variable(s) A description of the NIH Stroke Scale is given in Appendix 11.1. Descriptions of MoCA, GDS and SF36 are given in Appendices 11.5., 11.6. and 11.7, respectively.

CT Perfusion Protocol Appendix 11.8.

9.5.4. Safety variables

Safety Endpoints:

* patient survival at Day 90
* stroke-related and neurological deaths
* Adverse Events recording
* symptomatic cerebral haemorrhage defined as any blood in the brain or intracranially associated with a clinical deterioration of ≥4 points of the NIHSS for which the haemorrhage has been identified as the dominating cause of the neurologic deterioration
* cerebral herniation rate and symptomatic oedema
* vital sign measurement

ELIGIBILITY:
Inclusion Criteria:

* Female or male inpatients.
* Age: ≥18 years.
* MRS ≤2
* Clinical diagnosis of ischemic stroke eligible for EVT.
* No contraindication to undergo CT-Perfusion
* Patient is willing to participate voluntarily and to sign a written patient informed consent. Informed consent will be obtained from each patient or the legally authorised representative or two independent physicians, according to the regulatory and legal requirements of israel.

Exclusion Criteria:

Brain Imaging

• Evidence of intracranial haemorrhage (ICH) on the CT-scan

General

* Participation in another therapeutic clinical trial 3 months before baseline
* Female patient of childbearing age must not be pregnant as proved by Beta-HGB negative testing.

Medical

* Platelet count of below 100x103/mm3
* Blood glucose <50
* Known haemorrhagic diathesis
* Manifest or recent severe or dangerous bleeding
* Known bacterial endocarditis, pericarditis
* Acute pancreatitis
* Documented ulcerative gastrointestinal disease during the last 3 months, oesophageal varices, arterial-aneurysm, arterial/venous malformation
* Neoplasm with increased bleeding risk
* Severe liver disease, including hepatic failure, cirrhosis, portal hypertension, oesaphageal varices) and active hepatitis
* Major surgery or significant trauma in past 3 months
* Multiple serious drug allergies
* Hypersensitivity or allergy to one of the components of the drug
* Severe renal impairment Psychiatric
* Chronic intoxication or chronic substance use disorder with pharmaceuticals, drugs, alcohol or industrial poisons

Neurological

* Epilepsy
* Symptoms suggestive of subarachnoid haemorrhage, even if the CT-scan is normal
* Known history of or suspected intracranial haemorrhage
* Suspected subarachnoid haemorrhage or condition after subarachnoid hemorrhage from aneurysm
* Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
* Haemorrhagic retinopathy, e.g. in diabetes (vision disturbances may indicate haemorrhagic retinopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 Days
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. A standardized interview also exists to try to reduce subjectivity or variability in score assignments. Ranges between 0-6

SECONDARY OUTCOMES:
NIH Stroke Scale (NIHSS) | 90 Days
  The NIHSS is a 15-item neurological examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ranges between 0-42
Glasgow Outcome Score | 90 days
  The Glasgow Outcome Scale (GOS) categorizes the outcomes of patients after traumatic brain injury, as follows: Death. Persistent vegetative state: Minimal responsiveness. Severe disability: Conscious but disabled; dependent on others for daily support
Geriatric Depression Scale (GDS) | 90 days
  The Geriatric Depression Scale (GDS) is a self-report measure of depression in older adults. Users respond in a "Yes/No" format. The GDS was originally developed as a 30-item instrument
Montreal Cognitive Assessment (MoCA) | 90 days
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
Short Form 36 Health Survey (SF36) | 90 days
  A 36-item short-form (SF-36) was constructed to survey health status in the Medical Outcomes Study. The SF-36 was designed for use in clinical practice and research, health policy evaluations, and general population surveys.

OTHER OUTCOMES:
Symptomatic Intracranial Hemorrhage | 90 Days
  symptomatic cerebral haemorrhage defined as any blood in the brain or intracranially associated with a clinical deterioration of ≥4 points of the NIHSS for which the haemorrhage has been identified as the dominating cause of the neurologic deterioration
Patient Survivial at Day 90 | 90 days
  Survivial
Stroke related and Neurological Death | 90 days
  Death rate related to Stroke or Neurological Death

CONTACTS AND LOCATIONS:
Overall Officials: Roni Eichel, M.D., Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No